CLINICAL TRIAL: NCT02390440
Title: Liposomal Bupivicaine (Exparel) for Pain Control During Care of Rib Fractures
Brief Title: Exparel for Pain Control During Care of Rib Fractures
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not obtain an IND.
Sponsor: Michael Moncure, MD (Other)
Responsible Party: Sponsor-Investigator, Michael Moncure, MD, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRA_IIT_Exparel_RibFractures
Record Dates: First submitted 2015-03-03; First posted 2015-03-17 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Pain
Keywords: Pain management; Exparel; Rib fracture
MeSH Terms: conditions — Pain; Agnosia; Rib Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EXPAREL (Experimental): single dose, 266mg (20mL) of EXPAREL injected to slowly infiltrate the soft tissue around the site of fracture
  Interventions: Drug: EXPAREL

INTERVENTIONS:
Drug: EXPAREL
  Other Names: Liposomal Bupivicaine

SUMMARY:
This study is looking at a novel therapy of numbing medication injected directly around the fracture site. The purpose of this study is to determine if the study medication, EXPAREL®, is a viable alternative to current therapies for rib fractures.

DETAILED DESCRIPTION:
Rib fractures are common in patients who have suffered a traumatic injury, occurring in about 10% of general injury cases and in about 30% of cases where the injury is directly to the chest. Usually caused by injury to the chest wall, rib fractures most often occur where the ribs bend and are most fragile. These kinds of injuries are commonly caused by motor vehicle collisions, falls, assault, industrial accidents, gunshots, or repetitive causes such as severe coughing or use-injury in athletes. With any of these types of injury, the first concern of the physician is to repair any immediate damage to the chest wall (such as penetrating wounds, air or blood in the chest cavity that compresses the lung(s), or fixing the broken ribs in place). Once these injuries are repaired and stabilized, the patient's care consists of controlling their pain and helping them recover normal breathing ability.

In patients who are not admitted to the hospital for care, usually with only 1 or 2 ribs broken, care is often pain control using over the counter medicines like Tylenol or Ibuprofen (called NSAIDS) or prescription medicines like hydrocodone (Vicodin®). The main concern during follow-up of these patients is full recovery of pain-free breathing ability. In patients who are admitted to the hospital for treatment, pneumonia is the most common complication associated with multiple broken ribs. Pneumonia occurs in anywhere from 15% to 30% of these patients. For long-acting pain control to help them breathe more easily, studies have shown that epidural analgesia (pain relieving drugs delivered through a thin tube called a catheter into the fluid surrounding the spinal cord) is preferable over opioids, whether given in pill form or through an IV. Additional studies have shown better results with epidural pain control compared to opioid or NSAID use. However, with all of these methods come risks and side effects.

Using oral NSAIDs can result in stomach irritation, kidney injury, or can interfere with the body's ability to form blood clots. Acetaminophen (Tylenol) has been shown to be toxic to the liver at higher doses. Opioid use can lower a person's breathing ability even while it reduces their pain, which is not wanted in patients already at higher risk for pneumonia. Epidural placement is a complex procedure, risks infection at the site of catheter insertion, can cause itching, and risks injury to both the spinal cord and the membrane surrounding it (the dura).

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older
* patients with three or more rib fractures occurring either unilaterally or bilaterally
* patients who are awake enough to assess pain severity

Exclusion Criteria:

* patients whose pain in other anatomical areas limit rib fracture pain assessment
* patients with a history of hypersensitivity or idiosyncratic reactions or intolerance to any local anesthetic, opioids, or ketorolac
* patients who abuse alcohol or other drug substances
* patients on chronic opioid therapy (taken an opioid 5 of the last 7 days)
* pregnant patients
* severe hepatic impairment
* persistent pain patients requiring 20mg oral morphine equivalent or greater in the 24 hour period prior to sustaining multiple rib fractures
* allergies to common agents used in Exparel (bupivacaine, liposome)
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pain relief (visual analog scale) | Change from Treatment to Hour 72
  pain relief as measured by visual analog scale and patient satisfaction survey, before and after drug administration

SECONDARY OUTCOMES:
Length of hospital stay post treatment | Up to 10 days, average length of stay expected to be 3 days
  count of days participant in hospital post treatment
opioid use | Change from Treatment to Hour 72
change in lung function as evidenced by use of incentive spirometry | Change from Treatment to Hour 72
  Changes will be measured by using incentive spirometry. The incentive spirometry device includes an indicator which measures sustained inhalation vacuum. Change between performance will be measured at treatment to hour 72.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Moncure, MD, FACS, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States